CLINICAL TRIAL: NCT06729489
Title: Gastrointestinal Endoscopic Findings in Children With Referactory Iron Deficiency Anemia
Brief Title: Endoscopy in Anemic Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed ElSayed Mohamed Mohamed, Principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-2410-10MS
Record Dates: First submitted 2024-11-21; First posted 2024-12-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: Refractory Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Gastroscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with referactory iron deficiency anemia (Experimental)
  Interventions: Procedure: Upper Endoscopy

INTERVENTIONS:
Procedure: Upper Endoscopy — Endoscopy in children with refractory iron deficiency anemia
  Other Names: Colonoscopy

SUMMARY:
Assess the role of Upper and lower gastrointestinal endoscopy in evaluation of refractory iron deficiency anemia in children

ELIGIBILITY:
Inclusion Criteria:

* children with iron deficiency anemia not responding to medical treatment for more than 6 weeks

Exclusion Criteria:

* children with iron deficiency anemia responding to medical treatment Children below 1 years and above 18 years old

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Endoscopic findings in children with referactory iron deficiency anemia | 6 months
  Diagnosis of potential gastrointestinal tract causes of bleeding and anemia in children by using endoscopy and occult blood in stool and CBC and Iron profile

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided